CLINICAL TRIAL: NCT00328354
Title: Mammography SPECT With Rotating Slant Hole Collimator
Status: Withdrawn | Type: Observational
Why Stopped: Ran out of time/ funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: R01 EB 0019-83 Mammography
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The goal is to conduct a pilot study to determine the feasibility of the clinical use of RMSSH SPECT imaging technology for breast imaging and to develop a standardized clinical protocol.

DETAILED DESCRIPTION:
The goal of this protocol is to develop and evaluate a novel SPECT imaging technique for imaging the breast using rotating multi-segment slant-hole (RMSSH) collimators. The motivation is the requirement of a low cost RMSSH collimator and a conventional Large-Field-Of-View (LFOV) camera. It is believed that RMSSH SPECT is particularly suitable for applications in breast imaging.

ELIGIBILITY:
Inclusion Criteria:

* Women seen at Johns Hopkins Avon Division of Breast Imaging who have been diagnosed with breast cancer.

Exclusion Criteria:

* Pregnant (or possibly pregnant)
* Lactating
* Unable to give consent
* Weights over 300 pounds
* Women who have already undergone definitive surgical treatment to their breast for breast cancer will not be eligible.

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women seen at Johns Hopkins Avon Division of Breast Imaging who have been diagnosed with breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tsui, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States